CLINICAL TRIAL: NCT06346665
Title: The Transplant Cohort of the German Center for Infection Research
Status: Recruiting | Type: Observational
Sponsor: Technical University of Munich (Other)
Collaborators: Hannover Medical School (Other); University Hospital Heidelberg (Other); Universität Tübingen (Other); Klinikum der Universität München (Unknown); Max von Pettenkofer-Institut München (Unknown); Nierenzentrum Heidelberg (Unknown); Helmholtz Centre for Infection Research (Other)
Responsible Party: Sponsor
Other Study IDs: DZIF Tx-Cohort
Record Dates: First submitted 2024-03-26; First posted 2024-04-04 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-03

CONDITIONS: Infections; Transplant Complication; Transplant Failure; Immunosuppression
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Blood (Serum, plasma, RNA-stabilized, purified PBMC, buffy coat) Stool Urine Buccal swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Medical data and biological samples obtained from transplant patients are collected and managed across Germany with the help of the DZIF Transplant Cohort. The data and samples form the basis of scientific studies which investigate the connections between numerous factors influencing an organ's susceptibility to infection and organ function.

DETAILED DESCRIPTION:
Infections in transplant recipients have a decisive impact on graft function and survival of the transplant recipient, but many issues are still poorly understood. For example, little is known about the long-term consequences of many infections on graft survival/function and graft- versus-host disease (GvHD), the role of individual susceptibility to bacterial, viral and fungal colonisation under immune suppression, the evolution of the antiviral T cell repertoire, the long- term impact of antiviral therapy on graft and patient survival or changes in the physiological microbiome that may have a bearing on colonisation with pathogenic microbes. Taking advantage of the fact that most of the university hospitals with sizeable transplantation programs in Germany are also DZIF partners, we will establish a large multicentre prospective observational cohort of transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Consent
* undergone transplantation of kidney, pancreas, liver, heart or stem cells

Exclusion Criteria:

* No consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients of any age who have received a kidney, pancreas, liver, heart or stem cell transplant at one of the listed partner centres
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Realisation of studies that focus on the the medical needs of transplant patients, particularly with regard to their susceptibility to infection | 10 years
  Provision of collected data and biosamples to research groups for the realisation of scientific studies with a number of resources that individual clinics could not provide on their own

CONTACTS AND LOCATIONS:
Locations (1):
- Technische Universität München, München, Germany

IPD SHARING:
Plan to Share IPD: Yes
The use of collected data and biosamples is possible on the basis of an application to the Scientific Steering Committee of the transplant cohort. Cooperations with members of the cohort are welcome
Supporting Information: Study Protocol, ICF
Time Frame: The use of resources is possible after successful review of the preliminary and main application to the transplant cohort by the internal Scientific Steering Committee and - depending on the study design - external reviewers
URL: https://www.dzif.de/en/working-group/transplant-cohort

REFERENCES:
- [Result] Karch A, Schindler D, Kuhn-Steven A, Blaser R, Kuhn KA, Sandmann L, Sommerer C, Guba M, Heemann U, Strohaker J, Glockner S, Mikolajczyk R, Busch DH, Schulz TF; for the Transplant Cohort of the German Center for Infection Research (DZIF Transplant Cohort) Consortium. The transplant cohort of the German center for infection research (DZIF Tx-Cohort): study design and baseline characteristics. Eur J Epidemiol. 2021 Feb;36(2):233-241. doi: 10.1007/s10654-020-00715-3. Epub 2021 Jan 25. PMID 33492549
- [Result] Sommerer C, Schroter I, Gruneberg K, Schindler D, Behnisch R, Morath C, Renders L, Heemann U, Schnitzler P, Melk A, Della Penna A, Nadalin S, Heeg K, Meuer S, Zeier M, Giese T; Transplant Cohort of the German Center for Infection Research (DZIF Transplant Cohort) Consortium. Incidences of Infectious Events in a Renal Transplant Cohort of the German Center of Infectious Diseases (DZIF). Open Forum Infect Dis. 2022 May 13;9(7):ofac243. doi: 10.1093/ofid/ofac243. eCollection 2022 Jul. PMID 35855001
- See also: Transplant Cohort Website of the DZIF — https://www.dzif.de/en/working-group/transplant-cohort